CLINICAL TRIAL: NCT02492555
Title: Is Relapse Rate Reduced by Home Monitoring of IBD Patients Tightly or on Demand by FC and Disease Activity?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 48121
Record Dates: First submitted 2015-06-23; First posted 2015-07-08 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Inflammatory Bowel Disease
Keywords: IBD; Telemedicine; At-home monitoring; Disease activity; fecal calprotectin
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Scheduled (SI) (Experimental): "Scheduled" means screening every 3rd month ( home FC and DA) plus when needed and upgrade of ususal treatment
  Interventions: Other: SI
- On Demand (OD) (Active Comparator): On "Demand" means screening of home FC and DA when the patients feel for it and upgrade of usual treatment
  Interventions: Other: OD

INTERVENTIONS:
Other: SI — A routine scheduled (SI) screening of FC and DA every 3rd month
  Arms: Scheduled (SI)
Other: OD — A screening of FC and DA on demand (OD)
  Arms: On Demand (OD)

SUMMARY:
The purpose of this study is to determine if the IBD patient doing home monitoring by web app's for disease activity (DA) and fecal calprotectin (FC) on demand (OD), compared with patients doing home monitoring scheduled interval combined with "on demand"(SI+OD) ( every 3.month).

Will home monitoring of DA and FC OD vs SI+OD reduce frequency of relapse in one year follow up? Is the frequent FC measurement in SI+OD test group predictive of an early recognition of relapse, and thus help change the naturel course of disease? Will home monitoring of DA and FC in OD vs SI+OD change the course of the disease in terms of disease activity, spread of the disease, hospitalizations and number of hospitalization days, required surgery and outpatient visits? Is there a difference in patients' compliance with treatment plan between OD vs SI+OD ? Is there difference in patients-adherence between OD vs SI+OD ?

DETAILED DESCRIPTION:
Detailed Description Among 2.500 IBD patients the investigators will consecutively from the Gastroenterology out-patient clinic at North Zealand University Hospital recruit in total 120 in the study.

At the out-patient consultation IBD patients will be informed about the project and the IBD eHealth nurse ensures that no exclusion criteria met by the patient.

Inclusion criteria: IBD patients in remission, SCCAI ≤ 2 (Simple Clinical Colitis Activity Index )) or HBI < 5 (Harvey & Bradshaw Activity Index ) or in mild to moderate disease activity ( SCCAI 3-4, HBI < 16) IBD patients who can read, speak and understand Danish IBD patients that can take advantage of the Internet and wireless network 18years or older.

Exclusion criteria: IBD patients with severe disease activity HB > 16 SCCAI ≥ 5 ) IBD patients with social, medical or psychological issues of a more complex character IBD patients with particularly complex issues such as drug and alcohol problems, severe mental / psychiatric disorders and / or serious social impact.

IBD patients who cannot attend due language barrier or cognitive disorder. Age less 18. When the patient has agreed to participate in the study, randomized to either OD or SI OD 3. Months (SI group):

Patients log in at www.noh.constant-care.dk at least once every 3rd months throughout the project period of 12 months. When the patient log in to the telemedicine platform following scoring must be filled out:

1. - Disease activity, respectively SCCAI or HBI.
2. - Quality of life assessment, in s - IBDQ every 3rd months.
3. - FACIT (Fatigue score)
4. - MARS ( Medical Adherence Rating Scale)

   * FC, fecal calprotectin mg / kg feces) with SMART phone, rapid home test. If the patients prefer to send the feces test, it will be tested in the Gastro unit lab. at the hospital with SMART phone.

The results of the scoring systems will appear to the health professionals and patients in a traffic light turning into red, yellow and green.

If the patient experiences a recurrence of the disease, it moves from green to either yellow or red area in the traffic graph, and patient will further be instructed to contact Gastro medical clinic project nurse for an early consultation and decision on further treatment initiative. This will also be indicated at the patient's website. If alarm symptoms occurs patients are instructed to contact the project nurse. Thus patients are treated in accordance to national and international guideline. By screening of the inflammation burden the decision is moving forward.

On Demand Group:

Patients log in on demand,detects disease activity, quality of life and FC at the start, and subsequently when needed and at the end of the study (12 months).

At relapse disease activity score and FC is settled and repeated no later than 7 days here after at remission a new DA and FC test should be performed to verify the remission.

Statistical considerations:

Randomization Suitable (N = 120) will be randomized to one of the test groups by sealed envelope principle.

Material size calculation:

A relapse last in median 18 days in patients with inflammatory bowel disease, but the variance is large (10-50 days). During one year of a prevalent IBD patient group 50 % of a patient population will experience a relapse. To assess whether fewer patients experience true "red" indicated by relapse via (TIBS) Feces Calprotectin (FC ) and disease activity in group 1 vs. Group 2 respectively, the sample size has been depicted from TIBS and a statistically significance ( α ) of 0.05 , and test force of ( β ) of 0.8 .

This means that there must be included 53 individuals in each group, which means that there must be included a total of 106. Thus the investigators have chosen to include 120 patients, 60 in each group in order to correct for a possible of small drop out in each group.

ELIGIBILITY:
Inclusion Criteria:

* IBD patients in remission, SCCAI ≤ 2 (Simple Clinical Colitis Activity Index )) or HBI < 5 (Harvey & Bradshaw Activity Index ) or in mild to moderate disease activity ( SCCAI 3-4, HBI < 16)
* IBD patients who can read, speak and understand Danish
* IBD patients that can take advantage of the Internet and wireless network 18 years or older

Exclusion Criteria:

* IBD patients with severe disease activity ( HB > 16 SCCAI ≥ 5 )
* IBD patients with social, medical or psychological issues of a more complex character
* IBD patients with particularly complex issues such as drug and alcohol problems, severe mental / psychiatric disorders and / or serious social impact.
* IBD patients who cannot attend due language barrier or cognitive disorder.
* Age less 18.
* When the patient has agreed to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-07; Primary Completion 2016-08 (Actual); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Total Inflammation Burden Scoring ( TIBS) | 1 year
  The outcome measure of TIBS (FC ( ELISA Smartphone test)and Disease Activity ( Simple Clical Colitis Activity Index or Harvey-Bradshaw Index) has been chosen as endpoint for comparing the two screening methods in relation to relapse rate

CONTACTS AND LOCATIONS:
Overall Officials: Pia Munkholm, MD, Principal Investigator — professor
Locations (1):
- North Zealands Hospital, Frederikssund, Capital Region, Denmark